CLINICAL TRIAL: NCT01815073
Title: A Study to Evaluate the Immunogenicity and Safety of Live Attenuated Varicella Vaccine Combined With Live Attenuated JE Vaccine
Brief Title: Immunogenicity and Safety of Live Attenuated Varicella Vaccine Combined With Live Attenuated JE Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changchun Keygen Biological Products Co., Ltd. (Other)
Collaborators: Guangdong Provincial Institute of Biological Products And Materia Medica (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCT02049715
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Japanese Encephalitis; Chickenpox
MeSH Terms: conditions — Encephalitis, Japanese; Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Live Attenuated Varicella Vaccine + Live Attenuated JE Vaccine (Experimental): use the left arm flank deltoid muscle adheres to stick cohere place the skin after 75% ethyl alcohol disinfection the hypodermic injection
  Interventions: Biological: Live Attenuated Varicella Vaccine + Live Attenuated JE Vaccine
- Live Attenuated Varicella Vaccine (Experimental): use the right arm flank deltoid muscle adheres to stick cohere place the skin after 75% ethyl alcohol disinfection the hypodermic injection
  Interventions: Biological: Live Attenuated Varicella Vaccine
- Live Attenuated JE Vaccine (Experimental): use the right arm flank deltoid muscle adheres to stick cohere place the skin after 75% ethyl alcohol disinfection the hypodermic injection
  Interventions: Biological: live attenuated JE vaccine

INTERVENTIONS:
Biological: Live Attenuated Varicella Vaccine + Live Attenuated JE Vaccine
  Arms: Live Attenuated Varicella Vaccine + Live Attenuated JE Vaccine
Biological: Live Attenuated Varicella Vaccine
  Arms: Live Attenuated Varicella Vaccine
Biological: live attenuated JE vaccine
  Arms: Live Attenuated JE Vaccine

SUMMARY:
The purpose of this study is to observe the occurrence of adverse events and seroconversion rate, geometric mean titres (GMTs) of live attenuated varicella vaccine，live attenuated JE vaccine and live attenuated varicella vaccine combined with live attenuated JE vaccine, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal acceptable representative is willing and able to understand the protocol requirements and provide informed consent
* Participant is aged ≥ 1 year to ≤ 3 years
* Participant without previous history of chickenpox, zoster and epidemic encephalitis B
* Subject and parent/guardian able to attend all scheduled visits and comply with all trial procedures
* Body temperature ≤ 37.5℃

Exclusion Criteria:

* Known allergy to any constituent of the vaccine
* Known acute illness, severe chronic disease, acute exacerbation of chronic disease and fever
* Known or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth
* Reported the history of allergies, convulsions, epilepsy, mental illness and brain disease and clear serious systemic reaction
* Failed to the Expanded Programme on Immunization(EPI)
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Plan to receive any vaccine in the 4 weeks following the trial vaccination
* Known bleeding disorder
* Receipt of whole blood, blood plasma or immunoglobulin in the 5 months preceding the trial vaccination
* Reported the history of acute illness had need systemic antibiotics or anti-viral treatment of infections in the 7 days preceding the trial vaccination
* An acute illness with or without fever (temperature ≥ 38.0℃) in the 3 days preceding enrollment in the trial
* Participation in any other interventional clinical trial
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the vaccine

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 497 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate and GMTs for live attenuated varicella vaccine, live attenuated JE vaccine and live attenuated varicella vaccine combined with live attenuated JE vaccine, respectively. | 35-42 days after vaccination

SECONDARY OUTCOMES:
Occurrence of adverse events. | within 30 days after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Huizhen, Master, Principal Investigator — Guangdong Center for Disease Prevention and Control
Locations (1):
- Guangzhou Haizhu District Center for Disease Control and Prevention, Guangzhou, Guangdong, China